CLINICAL TRIAL: NCT01316991
Title: Understanding the Role of Chewing Gum in Satiation, Satiety and Hunger Management
Brief Title: A Study of Chewing Gum, Snacking and Appetite
Acronym: GUM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Nutrition Research Center, Illinois Institute of Technology (Industry)
Collaborators: Wm. Wrigley Jr. Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: GUM 2010-066
Record Dates: First submitted 2011-03-15; First posted 2011-03-16 (Estimated); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Hunger
Keywords: chewing gum; appetite; hunger; satiety; metabolic; nutrition; gut peptide hormones; psychological phenomena and processes
MeSH Terms: interventions — Chewing Gum

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chewing gum (Active Comparator): Subject will chew gum at defined intervals
  Interventions: Dietary Supplement: Chewing Gum
- No Gum (Placebo Comparator): No chewing gum will be provided to subject
  Interventions: Dietary Supplement: No Gum

INTERVENTIONS:
Dietary Supplement: Chewing Gum — chewing gum will be provided
  Other Names: subject will chew gum
  Arms: Chewing gum
Dietary Supplement: No Gum — no chewing gum will be provided
  Other Names: subject will not chew gum
  Arms: No Gum

SUMMARY:
Investigators are interested in learning how appetite responds after chewing gum.

In this research study subjects will be asked to eat a lunch meal provided at our Center. After eating the lunch meal, subjects will answer questions describing their feelings of hunger, thirst and desire to eat every 30 minutes for 3 hours.

Blood will be drawn throughout the study period to determine how chewing gum impacts certain hormones released from your intestine after eating and therefore how they influence your appetite. Blood draws will be done every 30 minutes for 3 hours. At only one of the two study visits, subjects will chew gum during specific times. One study visit will not include chewing gum.

After three hours, there will be a snack to eat as much as desired followed by one more set of questions and blood draw.

All study visits will take approximately 4 ½ hours.

DETAILED DESCRIPTION:
The study is a randomized, 2-arm, placebo-controlled, within-subjects crossover study to evaluate the satiety and metabolic response patterns of gum/no gum in relatively healthy weight and obese women.

The study will require one initial screening visit (1 hour) and 2 study visits. We are looking for healthy, non-smoking women older than 18 years of age with no significant medical history.

The initial screening visit will determine subject eligibility through height, weight and waist circumference measurements, vital signs, blood glucose test (finger prick) and completion of a series of surveys related to eating, health, exercise and mood.

If willing and eligible to participate, subjects will have 2 study visits. The lunch will be provided 4 hours after a intra-subject standardized breakfast (the same breakfast for each subject before each study visit). Upon arrival at each visit, subjects will have anthropometric measurements, vital signs upon blood glucose finger prick as well as assessment for compliance with breakfast protocol, subsequent fasting and adequate water intake.

Upon completion of pre-study procedures, a registered nurse will place a catheter (flexible tubing) in the subjects' arm during each study visit. A catheter is used so subjects are not stuck with a needle for every blood sample. Instead, the catheter is inserted using a needle, the needle is removed and the flexible plastic tubing remains the arm for the duration of the study day serving as a port for collecting blood samples at the specific time points

The initial blood draw will be collected (pre-lunch) then the lunch meal served. Subjects will have 20 minutes to finish the entire lunch meal. Thereafter, subjects will describe feelings of hunger, thirst and desire to eat every 30 minutes for 3 hours followed by blood draws.

At one of the 2 study visits, subjects will be provided chewing gum at which they will chew gum for 15 minutes leading up to the question set and blood draw.

A tray of snacks will be provided at 3 hours post-lunch and subjects may consume the snacks as desired. Lastly, a final set of questions will be answered followed by a blood draw at 4 hours post-lunch.

During the course of the study, subjects will be instructed to maintain their usual level of activity and a self-selected diet. Three day food records will be maintained throughout the course of the study.

Each study visit will last approximately 4 1/2 hours and subjects will be required to remain at the Clinical Nutrition Research Center on the IIT Campus for the duration of the visit.

ELIGIBILITY:
Inclusion Criteria:

* Females
* 18 years of age and older
* Healthy weight: BMI between 18.5 and 24.9 kg/m2, inclusive
* Obese: BMI between 30 - 38 kg/m2, inclusive
* No clinical evidence of cardiovascular, metabolic, respiratory, renal, gastrointestinal or hepatic disease
* Unrestrained eater (score < 10 on the Three Factor Eating Questionnaire)

Exclusion Criteria:

* Pregnant and/or lactating or planning for pregnancy
* Allergies or intolerances to foods consumed in the study
* Fasting blood glucose > 110 mg/dL. Subjects identified with elevated fasting blood glucose levels will be will be advised to contact their primary care physician for appropriate follow-up care.
* Taking over the counter supplements that may interfere with the study procedures or endpoints
* Taking prescription medications that may interfere with study procedures or endpoints (medications that affect appetite, unstable dose of hormones <6 months)
* Subjects with unusual dietary habits (e.g. pica)
* Actively losing weight or trying to lose weight (unstable body weight fluctuations of > 5 kg in a 60 day period)
* Excessive exercisers or trained athletes
* Addicted to drugs and/or alcohol
* Medically documented psychiatric or neurological disturbances
* Smoker (past smoker may be allowed if cessation is > 2 years)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2010-12-01 (Actual); Primary Completion 2015-09-01 (Actual); Study Completion 2015-09-01 (Actual)

PRIMARY OUTCOMES:
To characterize the subjective and metabolic satiety response pattern to chewing gum vs. no chewing gum on subjective satiety and subsequent second meal intake in adult women. | 4 hour post prandial study
  Chewing gum will be provided throughout the 4 hour post-prandial study at defined intervals at one of the two study visits. Feelings of hunger, fullness and desire to eat will be measured by the subject every 30 minutes post-lunch for 3 hours. Blood draws will also be collected every 30 minutes post-lunch for 3 hours.
  At 3 hours, a snack tray will be provided and subject will be instructed to consume as desired. One additional sent of questions and blood draw will be completed at 4 hours post-lunch.

SECONDARY OUTCOMES:
To investigate the relationship of metabolic responses to gum-induced/enhanced satiety by evaluating changes in free-living food intake in adult women | 2 days
  Blood draws will also be collected every 30 minutes post-lunch for 3 hours. One additional blood draw will be completed at 4 hours post-lunch.
  Subjects will be asked to maintain a self-selected diet throughout the study period. Leading up to the study visits, subjects will measure and record all food intake using food intake scales provided. Subjects will also be asked to measure and record all food intake for the remainder of the study visit day.

CONTACTS AND LOCATIONS:
Overall Officials: Britt Burton-Freeman, MS, PhD, Study Director — National Center Food Safety and Technology
Locations (1):
- Clinical Nutrition Research Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park E, Edirisinghe I, Inui T, Kergoat S, Kelley M, Burton-Freeman B. Short-term effects of chewing gum on satiety and afternoon snack intake in healthy weight and obese women. Physiol Behav. 2016 May 15;159:64-71. doi: 10.1016/j.physbeh.2016.03.002. Epub 2016 Mar 3. PMID 26948161